CLINICAL TRIAL: NCT00680459
Title: Ethanol Locks for the Treatment of Central Venous Line Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: inability to enroll adequate number of patients
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, christine mckiernan, Division Chief, Pediatric Critical Care, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB08-064
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-01

CONDITIONS: Bloodstream Infection
Keywords: central line infection; 70% ethanol; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Ethanol; Anticoagulants

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 70% ethanol lock solution instilled into central venous line of patient with documented infection, in addition to usual care with antimicrobials and supportive therapy. 70% ethanol solution dwells for 4 hours, then is withdrawn and discarded. This procedure repeated daily for 5 consecutive days.
  Interventions: Drug: 70% ethanol
- 2 (Placebo Comparator): heparin flush 10 units/ml lock solution instilled into central venous line of patient with documented infection, in addition to usual care with antimicrobials and supportive therapy. heparin flush solution dwells for 4 hours, then is withdrawn and discarded. This procedure repeated daily for 5 consecutive days.
  Interventions: Drug: heparin flush solution

INTERVENTIONS:
Drug: 70% ethanol — 70% ethanol lock solution instilled into central venous line of patient with documented infection, in addition to usual care with antimicrobials and supportive therapy. Volume of solution instilled varies from 0.8-1.9ml depending on volume of the lumen and hub of the particular size line being treated. 70% ethanol solution dwells for 4 hours, then is withdrawn and discarded. This procedure repeated daily for 5 consecutive days.
  Other Names: alcohol
  Arms: 1
Drug: heparin flush solution — heparin flush (10 units/ml) lock solution instilled into central venous line of patient with documented infection, in addition to usual care with antimicrobials and supportive therapy. Volume of solution instilled varies from 0.8-1.9ml depending on volume of the lumen and hub of the particular size line being treated. Heparin lock solution dwells for 4 hours, then is withdrawn and discarded. This procedure repeated daily for 5 consecutive days.
  Other Names: anticoagulant
  Arms: 2

SUMMARY:
Ethanol Locks as an Adjunct Treatment for Central Venous Line Infections

Purpose To evaluate the effectiveness of a 70% ethanol lock solution when used as an adjunct therapy with antibiotics to treat central venous line infections

Study Design Randomized Controlled Trial

Study Protocol Only those patients meeting all inclusion criteria and no exclusion criteria will be eligible to participate in this study. Once identified, signed informed consent will be obtained from the patient's guardian and the patient himself/herself depending on age. Patients will be randomized into 2 groups: Group 1 - those patients who will receive ethanol lock therapy and Group 2- those patients who will receive placebo therapy in the form of a heparin lock solution.

Outcome Measures Treatment success as defined by-

* Clearance of the infection as documented by negative blood cultures on day 6 (one day after completed of lock treatment)
* Preservation of the line at 30 days post treatment (day 35 of the study), this will be documented by a chart review in CIS and telephone interview to ensure no further growth from blood cultures or infections

Treatment failure as defined by-

* Clinical worsening during treatment
* Removal of the line due to persistent infection or sepsis
* Recurrence of infection with the same pathogen within 30 days

DETAILED DESCRIPTION:
Ethanol Lock Technique Protocol (adapted from the Children's Hospital Los Angeles)

1. Obtain a 3ml syringe made by the Baystate Pharmacy which will contain either sterile 70% ethanol solution or 10 units/ml heparin flush solution. Randomization into study groups will be performed by the pharmacy in patient blocks of 10. Treating physician and nurses will be blinded to patient group assignment. Syringes will be labeled "70% ethanol/heparin lock Study Solution"
2. Cleanse Hands
3. Use aseptic Technique throughout procedure
4. Clean injection cap/posi-flow cap with alcohol for 30 seconds and let dry
5. Unclamp the catheter and gently flush with normal saline to ensure patency of the catheter
6. Instill ethanol/heparin lock into the catheter to fill volume

   * Broviac Single Lumen 4.2 Fr (ID 0.7) Dose 0.8ml
   * Broviac Single Lumen 6.6 Fr (ID 1mm) Dose 0.8ml
   * Med-comp Single Lumen Catheter Dose 1.2ml
   * Hickman Double Lumen 7 Fr Distal (ID 1mm) Dose 1.2ml
   * Hickman Double Lumen 9 Fr Proximal (ID 0.7) Dose 1.2ml
   * Med-comp Double Lumen 8 or 10 Fr Dose 1.2ml
   * Port-a-cath- Any Port (including priming tubing) Dose 1.9ml
7. Clamp the catheter
8. Label the locked lumen with the provided label so that med is not flushed through the catheter
9. Let ethanol dwell in catheter continuously for 4 hours
10. When ethanol has dwelled for 4 hours, withdraw and discard the lock solution
11. The above procedure should be repeated daily for 5 consecutive days
12. The above procedure should be repeated to each lumen of the central venous catheter daily if there are multiple lumens

ELIGIBILITY:
Inclusion Criteria:

* age 6 months-23 years
* documented central line infection with bacteria or fungus (positive blood culture)

Exclusion Criteria:

* allergy or intolerance to ethanol
* pregnant or breastfeeding
* central line tunnel or exit site infection

Ages: 6 Months to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A McKiernan, MD, Principal Investigator — Baystate Medical Center; Amanda Conti, MD, Study Director — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Background] Onland W, Shin CE, Fustar S, Rushing T, Wong WY. Ethanol-lock technique for persistent bacteremia of long-term intravascular devices in pediatric patients. Arch Pediatr Adolesc Med. 2006 Oct;160(10):1049-53. doi: 10.1001/archpedi.160.10.1049. PMID 17018464

RESULTS

PARTICIPANT FLOW:
Groups:
- 70% Ethanol Solution: 70% ethanol lock solution instilled into central venous line of patient with documented infection, in addition to usual care with antimicrobials and supportive therapy. 70% ethanol solution dwells for 4 hours, then is withdrawn and discarded. This procedure repeated daily for 5 consecutive days.
- Heparin Flush: heparin flush 10 units/ml lock solution instilled into central venous line of patient with documented infection, in addition to usual care with antimicrobials and supportive therapy. heparin flush solution dwells for 4 hours, then is withdrawn and discarded. This procedure repeated daily for 5 consecutive days.
Period: Overall Study
Arm/Group | 70% Ethanol Solution | Heparin Flush
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 70% Ethanol Solution | Heparin Flush | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 13
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.4 (4.96) | 6.33 (4.0) | 6.9 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Clearance of Central Venous Line Infection by Day 6 of Study
Time Frame: 6 days
Measure: Number; unit: number of CVL cleared
Arm/Group | 70% Ethanol Solution | Heparin Flush
Number analyzed (Participants) | 7 | 6
number of CVL cleared | 7 | 6

2. Secondary Outcome: Preservation of Central Venous Line (Line Not Requiring Removal) by Day 35 of Study
Time Frame: 35 days
Measure: Number; unit: number of lines preserved
Arm/Group | 70% Ethanol Solution | Heparin Flush
Number analyzed (Participants) | 7 | 6
number of lines preserved | 6 | 6

3. Secondary Outcome: Recurrence of Central Venous Line Infection Within 35 Days of Enrollment
Time Frame: 35 days
Measure: Number; unit: # of pts with recurrent infection
Arm/Group | 70% Ethanol Solution | Heparin Flush
Number analyzed (Participants) | 7 | 6
# of pts with recurrent infection | 3 | 1

ADVERSE EVENTS:
Arm/Group | 70% Ethanol Solution | Heparin Flush
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No